CLINICAL TRIAL: NCT00190281
Title: Contrast-Enhanced US of Spleen, Liver and Kidney in Patients With Acute Infection (Malaria and Other Infectious Diseases: a Functional Study
Brief Title: Contrast-Enhanced US of Spleen, Liver and Kidney
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Other Study IDs: 04 025
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2005-03

CONDITIONS: Malaria; Pyelonephritis; Bacterial Infections
Keywords: FUNCTIONAL STUDY; CONTRAST-ENHANCED US; PERFUSION
MeSH Terms: conditions — Malaria; Pyelonephritis; Bacterial Infections

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
To evaluate the changes in the microcirculation of the liver, kidney and spleen during acute infection in patients with malaria (cohorts 1 and 3) and other infectious diseases such as acute pyelonephritis at day 0 (within 8 hours of the treatment start), day 2 to 4 and day 28-32, using functional US with continuous infusion of a contrast agent (SonoVue, Bracco, Italy).

Study hypothesis: malaria patients should exhibit a different pattern of enhancement, particularly when quantitative measurements of the SU signals is performed with destruction reperfusion kinetics.

DETAILED DESCRIPTION:
To evaluate the changes in the microcirculation of the liver, kidney and spleen during acute infection in patients with malaria (cohorts 1 and 3) and other infectious diseases such as acute pyelonephritis at day 0 (within 8 hours of the treatment start), day 2 to 4 and day 28-32, using functional US with continuous infusion of a contrast agent (SonoVue, Bracco, Italy).

Three cohortes will be studied: cohorte 1 infection at Plasmodium falciparum (24 patients), cohorte 3 infection at Plasmodium vivax, ovale or malariae (5 patients) and cohorte 2 other infectious diseases such as acute pyelonephritis (24 patients).

Study hypothesis: malaria patients should exhibit a different pattern of enhancement, particularly when quantitative measurements of the SU signals is performed with destruction reperfusion kinetics.

ELIGIBILITY:
Inclusion Criteria:

* Social security number
* Age over 18
* acute malaria infection or other infectious diseases
* Inpatients
* Signed informed consent form

Exclusion Criteria:

* Pregnancy
* Criteria of bad tolerance of infection
* Treatment started for more than 8 hours
* Lack of cooperation
* History of splenectomy, hematological disease, cirrhosis with portal hypertension, splenomegaly
* Medical treatment with beta blocker, diuretic, immunodepression drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53
Dates: Start 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Correas, MD PhD, Principal Investigator — NECKER UNIVERSITY HOSPITAL; Pierre Buffet, MD PhD, Study Director — Centre Médical - Institut Pasteur; Olivier Lortholary, MD PhD, Study Director — NECKER UNIVERSITY HOSPITAL
Locations (1):
- Department of Adult Radiology, Necker University Hospital, Paris, Île-de-France Region, France